

Sample size was determined with G\*power3 based on the results from pilot data of 0, 3 and 10 min stair climbing bouts (32 steps up and down) at self-selected stepping rate following consumption of a 75 g glucose drink. Specifically, with an effect size of  $\eta$  p2 = .144 and average correlation among repeated measures for the glucose area under curve of r = -.26 we calculated that a total sample size of N = 22 would be necessary to achieve power (1-  $\beta$  )  $\geq$  80% at the predetermined  $\alpha$ . Allowing for an attrition rate of 25% we will enroll a total of 30 participants.

Data will be analyzed with a 4 way repeated measures analysis of variance. The Level of significance will be set a priori at  $\alpha \le .05$